CLINICAL TRIAL: NCT01607138
Title: Speech and Swallowing Characteristics of Patients After Laryngectomy and the Effect on Quality of Life
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-12-CTJ-224-CTIL
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Cancer of the Larynx
Keywords: laryngectomy; swallowing disturbances; speech disturbances; speech intelligibility; voice prothesis
MeSH Terms: conditions — Laryngeal Neoplasms; Speech Disorders; Speech Intelligibility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total laryngectomy: A group of patients who underwent total laryngectomy with trechea esophageal puncture (TEP)

SUMMARY:
Swallowing and speech difficulties will be observed in patients post laryngectomy. These difficulties will cause decreased in quality of life.

DETAILED DESCRIPTION:
This study will explore the characteristics of speech and swallowing problems of patients who underwent laryngectomy.The relationship between swallowing disturbances and speech difficulties will be studied and the effect of each problem on quality of life will be messured.

ELIGIBILITY:
Inclusion Criteria:

* patients post total laryngectomy with voice prothesis

Exclusion Criteria:

* patients who can not read and respod to questions

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 adult patients, ages 35-80 y/o who underwent total laryngectomy and a trechea esophageal puncture was performed for the use of voice prothesis.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Speech and swallowing characteristics of patients post laryngectomy | At the completion of data collection -1 year
  After recording the patients' speech the speech characteristics will be analysed according to specific parameters. Also after performing swallowing eveluation swallowing disturbances will be diagnosed and described.

SECONDARY OUTCOMES:
The relationship between speech and swallowing disturbances of patients post laryngectomy | 1 year at the completion of data collection
  After analyzing the speech and swallowing disturbances of patients post laryngectomy, the relationship between these variables will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob T Cohen, PhD, Principal Investigator — Tel Aviv Medical Center

REFERENCES:
- [Background] * Maclean, J., Cotton, S., & Perry, A. (2009). Post-laryngectomy: it's hard to swallow: an Australian study of prevalence and self-reports of swallowing function after a total laryngectomy. Dysphagia, 24(2), 172-179. * Maclean, J., Cotton, S., & Perry, A. (2009). Dysphagia following a total laryngectomy: the effect on quality of life, functioning, and psychological well-being. Dysphagia, 24(3), 314-321. * McHorney, C. A., Robbins, J., Lomax, K., Rosenbek, J. C., Chignell, K., Kramer, A. E., & Bricker, D. E. (2002). The SWAL-QOL and SWAL-CARE outcomes tool for oropharyngeal dysphagia in adults: III. Documentation of reliability and validity. Dysphagia, 17(2), 97-114. * Platteaux, N., Dirix, P., Dejaeger, E., & Nuyts, S. (2010). Dysphagia in head and neck cancer patients treated with chemoradiotherapy. Dysphagia, 25(2), 139-152. * Kapila,M., Deore,N., Palav,R.S., Kazi,R.A., Shah,R.P., & Jagade,M.V.(2011). A brief review of voice restoration following total laryngectomy. Indian Journal of Cancer,48(1),99-104. * Rizzo,B.p.,Maronato,F.,Marchiori,C., Gava,A., &Da Mosto, M,C.(2008). Long-Term Quality of Life After Total Laryngectomy and Postoperative Radiotherapy Versus Concurrent Chemoradiotherapy for Laryngeal Preservation. The Laryngoscope.118,300-306 (2010). Total Laryngectomy.OtorhinolaryngologyMohebati,A. Mohebati,A & * Shah ,p .j , International Journal, 2(3), pp 207-214